CLINICAL TRIAL: NCT04685616
Title: A Randomised Phase III Trial With a PET Response Adapted Design Comparing ABVD +/- ISRT With A2VD +/- ISRT in Patients With Previously Untreated Stage IA/IIA Hodgkin Lymphoma
Brief Title: Brentuximab Vedotin in Early Stage Hodgkin Lymphoma
Acronym: RADAR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Takeda (Industry); University of Miami (Other); European Organisation for Research and Treatment of Cancer - EORTC (Network); Australasian Leukaemia and Lymphoma Group (Other); Seagen Inc. (Industry); Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RADAR; 2020-005160-65 (EudraCT Number); IISR X25041 (Other Grant/Funding Number: Takeda Pharmaceutical Company Ltd); UCL/15/0105 (Other: UCL); CCTG HD.12 (Other: CCTG); IRB number 20230081 (Other: University of Miami)
Record Dates: First submitted 2020-11-27; First posted 2020-12-28 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-05

CONDITIONS: Hodgkin Lymphoma
Keywords: PET-response adapted; Stage IA/IIA Hodgkin lymphoma; Brentuximab vedotin
MeSH Terms: conditions — Hodgkin Disease | interventions — Doxorubicin; Bleomycin; Brentuximab Vedotin; Vinblastine; Dacarbazine; Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABVD +/- ISRT (Active Comparator): 2 x 28 day cycles of ABVD: Doxorubicin 25mg/m^2 IV days 1 & 15 Bleomycin 10000 IU/m^2 days 1 & 15 Vinblastine 6mg/m^2 days 1 & 15 Dacarbazine 375mg/m^2 days 1 & 15
  PET-CT after 2 cycles will determine subsequent treatment:
  Deauville score 1-3 (PET CMR): 1 further cycle of ABVD then follow up Deauville score 4 (PET positive): 2 further cycles of ABVD followed by involved site radiotherapy (ISRT) Deauville score 5: withdraw from trial treatment; further treatment will be given at the treating clinician's discretion. Enter follow up for the trial.
  Interventions: Radiation: Involved site radiotherapy; Drug: Doxorubicin; Drug: Bleomycin; Drug: Vinblastine; Drug: Dacarbazine
- A2VD +/- ISRT (Experimental): 2 x 28 day cycles of A2VD: Doxorubicin 25mg/m^2 IV days 1 & 15 Brentuximab vedotin 1.2mg/kg (max 120mg) days 1 & 15 Vinblastine 6mg/m^2 days 1 & 15 Dacarbazine 375mg/m^2 days 1 & 15 Filgrastim (or equivalent haematopoietic growth factor) for 5-7 days from day 2 and day 16 (or single dose of peg-filgrastim on days 2 & 16)
  PET-CT after 2 cycles will determine subsequent treatment:
  Deauville score 1-3 (PET CMR): 1 further cycle of A2VD then follow up Deauville score 4 (PET positive): 2 further cycles of A2VD followed by involved site radiotherapy (ISRT) Deauville score 5: withdraw from trial treatment; further treatment will be given at the treating clinician's discretion. Enter follow up for the trial.
  Interventions: Radiation: Involved site radiotherapy; Drug: Doxorubicin; Drug: Brentuximab vedotin; Drug: Vinblastine; Drug: Dacarbazine; Drug: Haematopoietic growth factor

INTERVENTIONS:
Radiation: Involved site radiotherapy — Involved site radiotherapy as per International Lymphoma Radiation Oncology Group (ILROG) guidelines.
  Recommended dose 30Gy
Drug: Doxorubicin — See arm description
Drug: Bleomycin — See arm description
  Arms: ABVD +/- ISRT
Drug: Brentuximab vedotin — See arm description
  Arms: A2VD +/- ISRT
Drug: Vinblastine — See arm description
Drug: Dacarbazine — See arm description
Drug: Haematopoietic growth factor — See arm description
  Other Names: Filgrastim; G-CSF; Pegfilgrastim
  Arms: A2VD +/- ISRT

SUMMARY:
RADAR is a multicentre, international, randomised, open-label phase III clinical trial composed of 2 trials running in parallel. Trial 1 will be led and sponsored by University College London (UCL) and conducted in Europe and Australia/New Zealand. Trial 2 will be led by the Canadian Cancer Trials Group (CCTG) and conducted in North America, with CCTG the regulatory sponsor in Canada, and University of Miami the regulatory sponsor and IND holder in the US. Datasets from Trial 1 and Trial 2 will be combined to achieve the total sample size. Data analysis will be performed by UCL and therefore UCL is responsible for the clinicaltrials.gov entry.

Eligible patients will be randomised to receive either ABVD or A2VD chemotherapy.

An interim PET-CT scan will be performed after 2 cycles of treatment, which will be used to adapt subsequent treatment. Patients will receive a total of 3-4 cycles of chemotherapy and may also receive involved site radiotherapy as consolidation.

Patients will be followed up for a minimum of 5 years after treatment.

DETAILED DESCRIPTION:
Eligible patients will be randomised to receive either ABVD chemotherapy (doxorubicin, bleomycin, vinblastine and dacarbazine) or A2VD chemotherapy (doxorubicin, brentuximab vedotin, vinblastine and dacarbazine, with growth factor support).

If patients agree, they will have a PET-CT scan after 1 cycle (PET1). The result of this scan will be blinded and used for exploratory endpoints only. Treatment will not be influenced by the result of this scan.

All patients will have a PET-CT scan after 2 cycles of treatment (PET2) which will be centrally reviewed. The Deauville score from central review will be used to risk adapt subsequent therapy as follows:

* Patients with Deauville score 1-3 will have one further cycle of their randomised chemotherapy and then enter follow up.
* Patients with Deauville score 4 will have two further cycles of their randomised chemotherapy followed by involved site radiotherapy
* Patients with Deauville score 5 will be withdrawn from trial treatment. They will have further treatment at their treating clinician's discretion and will enter follow up for the trial.

Patients with Deauville score 4 on PET2 will have a final PET-CT scan to confirm adequate treatment response.

Patients will be followed up for a minimum of 5 years after completing treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 16-69 years (inclusive) (age range is 18-69 in US and EU)
* Histologically confirmed classical Hodgkin lymphoma
* Stage I or II supradiaphragmatic disease with no mediastinal bulk disease (defined as greater than a third of the transthoracic diameter at any level of thoracic vertebra as determined by CT) or B symptoms. Bulky disease at other sites is acceptable. Extranodal disease (single extranodal site (stage I) or contiguous nodal extension (stage II)) is acceptable.
* ECOG performance status 0-2.
* No previous treatment for Hodgkin lymphoma
* Fit to receive anthracycline-based chemotherapy (patients with a history of ischaemic heart disease or hypertension should have a left ventricular ejection fraction of ≥50%)
* Creatinine clearance (measured or calculated >40ml/min
* Total bilirubin <1.5 x upper limit of normal, unless attributable to disease or known Gilbert's syndrome
* ALT or AST < 2 x upper limit of normal
* Adequate bone marrow function with neutrophils ≥1.0x10^9/l and platelets ≥100x10^9/l
* Haemoglobin ≥8g/dL
* Willing and able to comply with the requirements of the protocol, including contraceptive advice, where applicable
* Written informed consent

Exclusion Criteria:

* Previous treatment for Hodgkin lymphoma, excluding short courses of oral corticosteroids at a dose of 100mg prednisolone (or equivalent) for up to 7 days
* Infradiaphragmatic disease
* Nodular lymphocyte predominant Hodgkin lymphoma
* Absence of FDG-avid lesions on baseline PET scan
* Age 70 years or over or age 15 years or under
* Other cancer diagnosed with the last 5 years. Patients with completely excised carcinoma in situ of any type and basal or squamous cell carcinoma of the skin are not excluded
* Recurrent or persistent other cancer within last 5 years irrespective of date of initial diagnosis
* Pre-existing grade ≥1 sensory or motor neuropathy from any cause
* History of or current progressive multi-focal leukoencephalopathy or other chronic condition of the brain
* Symptomatic neurologic disease compromising normal activities of daily living or requiring medications
* Infection with HIV, hepatitis C or active hepatitis B infection (surface antigen or DNA positive)
* Any active systemic viral, bacterial or fungal infection requiring systemic antibiotics, antivirals or antifungals within 2 weeks prior to first trial drug dose
* Receiving or recently treated with any other investigational agent (within 4 weeks of trial entry)
* Pregnant or breastfeeding women
* Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin or any component of ABVD
* Known history of any cardiovascular or respiratory conditions that would preclude anthracycline or bleomycin administration
* Other significant medical or psychiatric comorbidity that in the opinion of the investigator would make administration of ABVD or A2VD hazardous

Ages: 16 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1042 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 3 years from end of treatment
  Time from randomisation to first date of progression or death

SECONDARY OUTCOMES:
PET-CMR (complete metabolic response) rate | At the end of cycle 2 (each cycle is 28 days)
  Proportion of patients who have Deauville score 1-3 on PET-CT scan
Event-free survival (EFS) | 5 years from end of treatment
  Time from randomisation to first date of progression, death or a positive PET2 scan (whichever occurs first)
Overall survival (OS) | 5 years from end of treatment
  Time from randomisation to death
Incidence of second cancers and cardiovascular disease | 5 years from end of treatment
  Proportion in each arm who develop a second cancer or cardiovascular disease
Safety and toxicity of ABVD and A2VD as described by CTCAE v5.0 | From start of treatment to 30 days post treatment
  Numbers of patients experiencing a grade 3+ adverse event of each type will be presented and compared between the arms. Only patients who start treatment will be included

OTHER OUTCOMES:
Prognostic power of PET after 1 and 2 cycles of ABVD/A2VD | Up to 5 years after end of treatment
  7A Associations between PET1 Deauville score (DS) and PET2 DS; 7B Associations between PET1 DS and EFS; 7C Associations between PET1 DS and OS; 7D Associations between PET1 DS and PFS; 7E Associations between PET2 DS and EFS; 7F Associations between PET2 DS and OS; 7G Associations between PET2 DS and PFS; 7H Associations between EORTC baseline stratification and PET1 DS; 7I Associations between EORTC baseline stratification and PET2 DS; 7J Associations between EORTC baseline stratification and EFS; 7K Associations between EORTC baseline stratification and OS; 7L Associations between EORTC baseline stratification and EFS; 7M Associations between GHSG baseline stratification and PET1 DS; 7N Associations between GHSG baseline stratification and PET2 DS; 7O Associations between GHSG baseline stratification and EFS; 7P Associations between GHSG baseline stratification and OS; 7Q Associations between GHSG baseline stratification and EFS
Prognostic and predictive power of baseline PET features | Up to 3 years after end of treatment
  The association of baseline quantitative PET parameters such as total lesion glycolysis (TLG) and PFS/EFS/OS will be assessed. The ability to predict PET score (PET1 and PET2) and Hodgkin lymphoma events within 3 years will be compared: 8A Associations between baseline quantitative PET parameters such as total lesion glycolysis (TLG) and PFS; 8B Associations between baseline quantitative PET parameters such as total lesion glycolysis (TLG) and OS; 8C Associations between baseline quantitative PET parameters such as total lesion glycolysis (TLG) and EFS; 8D Associations between baseline quantitative PET parameters such as total lesion glycolysis (TLG) and PET1 DS; 8E Associations between baseline quantitative PET parameters such as total lesion glycolysis (TLG) and PET2 DS
Change in pulmonary function tests at end of treatment, 1 and 2 years | 3 months & 1 year after end of treatment
  Change from baseline pulmonary function test (DLCO/TLCO percentage of normal) will be compared
Correlation between maximum tumour dimension at baseline and end of treatment with PFS | Up to 5 years after end of treatment
  The relationship between maximum tumour dimension at baseline and at end of treatment and PFS will be examined. This may also be analysed within the groups that achieve/do not achieve CMR after 2 cycles and may also be adjusted for the use of consolidation radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: John Radford, Principal Investigator — University of Manchester / Christie Hospital, Manchester
Locations (65):
- United States (3):
  - Stanford University - (Stanford Cancer Institute), Stanford, California
  - University of Miami School of Medicine, Miami, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Australia (10):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Townsville University Hospital, Townsville, Queensland
  - Royal Adelaide Hospital, Adelaide
  - Box Hill Hospital, Box Hill
  - Royal Brisbane and Women's Hospital, Brisbane
  - Royal Darwin Hospital, Darwin
  - Liverpool Hospital, Liverpool
  - Sunshine Hospital (Western Health), Melbourne
  - Concord Repatriation General Hospital, Sydney
  - St George Hospital, Sydney
- Belgium (4):
  - AZ Delta Campus Rumbeke, Roeselare, West Flanders
  - Ziekenhuis Netwerk Antwerpen, Antwerp
  - UZ Leuven, Leuven
  - CHU-UCL Namur, Namur
- Canada (6):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Ottowa Hospital Research Institute, Ottawa
  - Saint John Regional Hospital, Saint John
  - University Health Network Princess Margaret Cancer Centre, Toronto
  - Vancouver Cancer Centre, Vancouver
  - CancerCare Manitoba, Winnipeg
- Denmark (2):
  - Aarhus University Hospitak Skjeby, Aarhus
  - Rigshospitalet, Copenhagen
- Netherlands (5):
  - Amsterdam UMC - location VUMC, Amsterdam
  - Reinier de Graafweg 3-11 - Postbus 5011 - 2625 AD Delft, Delft
  - Universitair Medisch Centrum Groningen, Groningen
  - Radboud University Medical Center Nijmegen, Nijmegen
  - NL 331 - Haaglanden Medisch Centrum (HMC) - Haaglanden MC, The Hague
- Auckland City Hospital, Auckland, New Zealand
- Instituto Portugues de Oncologia de Lisboa Francisco Gentil, Lisbon, Portugal
- Narodny Onkologicky Ustav, Bratislava, Slovakia
- Spain (3):
  - Hospital Del Mar, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - Complejo Hospitalario de Navarra, Pamplona
- United Kingdom (29):
  - University Hospital of Wales, Cardiff & Vale University Local Health Board, Cardiff, Cardiff
  - Blackpool Victoria Hospital, Blackpool, Lancashire
  - Freeman Hospital, Newcastle, Newcastle upon Tyne, Newcastle
  - Nottingham University Hospitals NHST, Nottingham, Nottingham
  - Lanarkshire, Glasgow, Scotland
  - St George's Hospital, London, Tooting
  - Aberdeen Royal Infirmary, Aberdeen
  - University Hospitals Birmingham, Birmingham
  - Glan Clwyd Hospital, Bodelwyddan
  - Bristol Haematology and Oncology Centre, Bristol
  - Colchester Hospital, ESNEFT, Colchester
  - University Hospital Coventry, Coventry
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Castle Hill Hospital, Hull
  - University Hospitals of Leicester NHS Trust, Leicester
  - The Clatterbridge Cancer Centre NHSFT, 65 Pembroke Place, Liverpool
  - St Bartholomew's Hospital, London
  - University College London Hospitals NHS Foundation Trust (UCLH), London
  - Royal Marsden Hospital Chelsea, London
  - Christie Hospital, Manchester
  - Norfolk & Norwich University Hospital, Norwich
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Royal Hallamshire Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Sunderland Royal Hospital, Sunderland
  - Royal Marsden Hospital, Sutton
  - Torbay Hospital, Torquay
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712